CLINICAL TRIAL: NCT05068271
Title: Effects of Multi-Domain Exercise Intervention on Memory Performance in Healthy Adults With and Without ApoE e4 Allele: A fMRI Study
Brief Title: Multi-Domain Exercise and Memory in Adults Relative to ApoE Genotype: A fMRI Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Kai Chang, Professor, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PACNL_WEBFIT: Memory & fMRI
Record Dates: First submitted 2021-07-19; First posted 2021-10-05 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Exercise Training; Executive Function; Aging
Keywords: multiple fitness; meditation; mindfulness; Apolipoprotein E; aging; magnetic resonance images; memory
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Domain Exercise Program (Experimental): Time: 6 months, total of 150 min of exercise per week.
  Intervention: aerobic training, muscular fitness training, balance, flexibility, meditation, and social interaction.
  Interventions: Behavioral: Multi-Domain Exercise Program
- Control Group (Other): Time: 6 months, total of 60 min of online educational course per week.
  Intervention: educational materials relating to the effects of exercise on cognitive function and aging-related cognitive decline.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Multi-Domain Exercise Program — The multi-domain exercise consisted of the main exercise (e.g., aerobic exercise, resistance exercise, flexibility training, and coordinative exercise), social interaction, and meditation. Participants are encouraged to engage in 150 min exercise per week consisting of one 90-min on-site session and multiple online sessions for 6 months.
  Arms: Multi-Domain Exercise Program
Behavioral: Control Group — The "usual physical activity group," as the control group, is informed to maintain their lifestyles. In addition, participants are invited to attend one 60-min online educational course per week. The logs of physical activity behavior will be obtained from the participants once per month during the intervention period.
  Arms: Control Group

SUMMARY:
The current project utilizes a single-blinded, double arm, 6-month randomized controlled trial to assess the effects of a multi-domain exercise program on memory performance, as well as cortical activities during the memory tasks in cognitively intact adults (i.e., 45-70 years). In addition, the potential moderator role of apolipoprotein epsilon-4 (ApoE e4) status and the mediator role of the brain-derived neurotrophic factor (BDNF) will be explored.

DETAILED DESCRIPTION:
Aging has been adversely associated with the deterioration of cognitive and brain functions. Most research on the effects of regular exercise on cognitive and brain functions has been focused on exercise programs with a single mode of exercise. Studies focusing on the effects of exercise programs with multi-domains on cognitive function and cortical functionality are sparse in late-middle-aged and older adults. In addition, while growing evidence has revealed the beneficial effects of regular exercise on cognitive function, scientific evidence regarding the effects of multi-domain exercise programs on cognitive function and brain function in late-middle-aged and older adults who are with or without the genetic risk for Alzheimer's disease (AD) is scarce. Lastly, the potential mediator role of the brain-derived neurotrophic factor (BDNF) in individuals is required to be explored.

In the current study, a single-blinded, double arm, 6-month randomized controlled trial has been utilized to assess the effects of a multi-domain exercise program containing multiple physical fitness components, meditation, and social interaction on memory, as well as cortical functionalities during the memory tasks in cognitively intact adults (i.e., 45-70 years). Specifically, the project aims to examine: (1) the causal links between a multi-domain exercise program composed of various physical fitness components, meditation, and social interaction against a control group on the memory performance in cognitively intact adults aged between 45 and 70 years with or without a genetic risk for AD, (2) the cortical functionality through functional images collected through a series of functional magnetic resonance images (fMRI), and (3) the potential influence of apolipoprotein epsilon-4 (ApoE e4) and BDNF on the effects of exercise.

One hundred eligible individuals will participate in the current study and will be randomly assigned into either the 6-month multi-domain exercise group (exercise group) or the online educational course group (control group).

All participants' physical fitness, cognitive function, and cortical functionalities via fMRI scanning will be assessed at the Baseline (Baseline-Assessments) and at the cessation of the 6-month intervention (Post-Assessments). The potential moderating role of ApoE genotypes and the mediation role of BDNF will be explored. Participation in this study will take approximately 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal vision
* Able to speak and read Chinese
* Scores of Mini-Mental Status Examination >= 25
* Physical Activity Readiness Questionnaire score < 0
* Able to conduct the exercise with moderate intensity
* Meet the criteria to undergo magnetic resonance imaging
* Provide informed consent

Exclusion Criteria:

* Diagnosed or self-reported cognitive problems (e.g., mild cognitive impairment or dementia)
* Diagnosed or self-reported physical disease (e.g., untreated hypertension and chronic heart disease, stroke, brain tumor, musculoskeletal disorders, other exercise contradictions)
* Diagnosed or self-reported major psychiatric illness (e.g., major depression, schizophrenia)
* Diagnosed or self-reported neurodegenerative disease (e.g., Alzheimer's disease and other dementias, Parkinson's disease (PD) and PD-related disorders, Huntington's disease)
* History of alcohol or drug abuse
* History of chemotherapy
* Traveling consecutively for three weeks or more during the study
* Unwillingness to be randomized to one of the two groups
* Currently participating in another study trial

Exclusion Criteria for functional magnetic resonance images (fMRI):

Participants will be excluded if s/he has a contraindication to fMRI scanning, such as aneurysm clip, implanted neural stimulator, cochlear implant, any implanted device, cardiac pacemaker. To ensure volunteers are eligible for the current project, they will be asked to fill out a questionnaire to inform whether they have conditions (e.g. paralyzed hemidiaphragm) or present unnecessary risks (e.g., pregnancy) during the recruitment period.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes in functional MRI indices | 60 min each at the Baseline-Assessment and at the Post-Assessment
  Functional MRI assessments will be conducted at the baseline (Baseline-Assessment) and at the end of the 6-month intervention (Post-Assessment) to measure participants' brain functionalities. Changes in functional MRI indices between the Baseline-Assessment and Post-Assessment will be assessed.
Changes in working memory performance: N-back working memory task | 30 min assessment time at the Baseline-Assessment and at the Post-Assessment
  Working memory performance will be assessed using the computerized n-back working memory task at the baseline (Baseline-Assessment) and at the end of the 6-month intervention (Post-Assessment). A total of 6 blocks with 108 trials (18 trials each block) will be utilized in the current study. Changes in working memory performance between the Baseline-Assessment and Post-Assessment will be assessed.
Changes in episodic memory performance: Relational and item-specific encoding and recognition test | 30 min each session at the Baseline-Assessment and at the Post-Assessment
  Episodic memory performance will be assessed using the relational and item-specific encoding and recognition test at the baseline (Baseline-Assessment) and at the end of the 6-month intervention (Post-Assessment). Changes in episodic memory performance between the Baseline-Assessment and Post-Assessment will be assessed.

SECONDARY OUTCOMES:
ApoE genotype | 5 min at the Baseline Assessment
  Based on the genetic biomarkers (rs429358 and rs7412), participants' ApoE genotype will be determined.
Changes in blood neurotrophic marker: Brain-derived neurotrophic factor (BDNF) | 5 min each at the Baseline-Assessment and at the Post-Assessment
  A 6 mL serum sample will be drawn from the antecubital vein at the baseline (Baseline-Assessment) and at the end of the 6-month intervention (Post-Assessment) to determine the concentration of BDNF. Changes in BDNF levels between the Baseline-Assessment and Post-Assessment will be assessed.
Physical fitness measurements: Changes in aerobic fitness | 20 min each at the Baseline-Assessment and at the Post-Assessment
  Participants' aerobic fitness will be estimated using the submaximal cycle ergometer test at the baseline (Baseline-Assessment) and at the end of the 6-month intervention (Post-Assessment). Changes in aerobic fitness between the Baseline-Assessment and Post-Assessment will be assessed.
Physical fitness measurements: Changes in muscular fitness | 15 min each at the Baseline-Assessment and at the Post-Assessment
  Muscular fitness will be assessed using either the push-up test/30sec or the chair stand test/30sec at the baseline (Baseline-Assessment) and the end of the 6-month intervention (Post-Assessment). A higher number completed indicated a better level of muscular fitness. Changes in muscular fitness between the Baseline-Assessment and Post-Assessment will be assessed.
Physical fitness measurements: Changes in flexibility | 15 min each at the Baseline-Assessment and at the Post-Assessment
  Flexibility will be assessed using the sit-and-reach test at the baseline (Baseline-Assessment) and at the end of the 6-month intervention (Post-Assessment). Further distance indicates better lower back and hip joint flexibility. Changes in flexibility between the Baseline-Assessment and Post-Assessment will be assessed.
Physical fitness measurements: Changes in body composition | 15 min each at the Baseline-Assessment and at the Post-Assessment
  The body composition (e.g., body water, body fat, skeletal muscle mass, body mass index, and percentage of body fat) will be assessed simultaneously using a body composition analyzer (ACCUNIQ BC380 Body Composition Analysis, SELVAS Healthcare Inc., Korea) at the baseline (Baseline-Assessment) and at the end of the 6-month intervention (Post-Assessment). Changes in body composition between the Baseline-Assessment and Post-Assessment will be assessed.
Psychosocial measures: Changes in mindfulness | 5 min each at the Baseline-Assessment and at the Post-Assessment
  Levels of mindfulness will be assessed using the 15-items (1-6 Likert scale) WHOQOL-OLD-Taiwan Chinese version of the Mindful Attention Awareness Scale questionnaire at the baseline (Baseline-Assessment) and at the end of the 6-month intervention (Post-Assessment). Higher scores are associated with higher dispositional mindfulness. Changes in mindfulness levels between the Baseline-Assessment and Post-Assessment will be assessed.
Psychosocial measures: Changes in sleep quality | 5 min each at the Baseline-Assessment and at the Post-Assessment
  Sleep quality is assessed by the Pittsburgh Sleep Quality Index. The questionnaire consists of 9 questions. Lower scores are associated with better sleep quality. Changes in sleep quality between the Baseline-Assessment and Post-Assessment will be assessed.
Psychosocial measures: Changes in depression | 5 min each at the Baseline-Assessment and at the Post-Assessment
  Depression level is assessed by the Chinese version of the Geriatric Depression Scale (GDS-15). The questionnaire consists of 15 'Yes/No' items. The total scores between 5 and 9 indicate mild symptoms, and a score of 10 and above indicates moderate symptoms. Changes in depression levels between the Baseline-Assessment and Post-Assessment will be assessed.
Psychosocial measures: Changes in health-related quality of life | 10 min each at the Baseline-Assessment and at the Post-Assessment
  Health-related quality of life is assessed by the 24-items (1-5 Likert scale) WHOQOL-OLD-Taiwan. The higher total scores indicate better quality of life. Changes in health-related quality of life between the Baseline-Assessment and Post-Assessment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, PhD, Principal Investigator — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (2):
- Taiwan (2):
  - Yu-Kai Chang, Taipei
  - National Taiwan Normal University, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang YK, Erickson KI, Aghjayan SL, Chen FT, Li RH, Shih JR, Chang SH, Huang CM, Chu CH. The multi-domain exercise intervention for memory and brain function in late middle-aged and older adults at risk for Alzheimer's disease: A protocol for Western-Eastern Brain Fitness Integration Training trial. Front Aging Neurosci. 2022 Aug 18;14:929789. doi: 10.3389/fnagi.2022.929789. eCollection 2022. PMID 36062144